CLINICAL TRIAL: NCT00918086
Title: Impact of Vitamin D Supplementation on Host Immunity to Mycobacterium Tuberculosis and Response to Treatment: Building Translational Research Capacity in Nutrition and Infectious Diseases in the Republic of Georgia
Brief Title: Impact of Vitamin D Supplementation on Host Immunity to Mycobacterium Tuberculosis and Response to Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Thomas R. Ziegler, MD, Professor of Medicine, Emory University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: IRB00014641; Vitamin D Georgia Study (Other: Other)
Record Dates: First submitted 2009-06-10; First posted 2009-06-11 (Estimated); Last update posted 2014-07-11 (Estimated); Status verified 2014-07

CONDITIONS: Tuberculosis
Keywords: Vitamin D; Tuberculosis
MeSH Terms: conditions — Tuberculosis | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin D pill (Experimental)
  Interventions: Dietary Supplement: Vitamin D pill
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D pill — Oral tablet taken for 16 weeks
  Arms: Vitamin D pill
Dietary Supplement: Placebo — An inactive pill that looks and tastes like the Vitamin D pill
  Arms: Placebo

SUMMARY:
Tuberculosis bacterium (TB) is a germ that can infect any part of the human body, especially the lungs. Vitamin D is a hormone present in humans that regulates blood electrolytes such as calcium and phosphate. There is new information that links vitamin D to the functioning of our immune system. The purpose of the study is to find out how vitamin D affects the immune system of patients with TB. We want to find out if correcting low vitamin D levels, in addition to getting standard therapy for TB, will help the immune system fight off TB infection more effectively.

The study will be done at the Georgia National Center for Tuberculosis and Lung Diseases (NCTBLD) in Tbilisi, Republic of Georgia. 220 patients with tuberculosis and 80 family members or household contacts of patients with tuberculosis will be participating in this study. TB patients, already receiving standard TB therapy, will be randomly assigned to either receive the Vitamin D pill or a placebo for a total of sixteen weeks. Neither the subject nor the investigator will know whether the subject has received the Vitamin D or the inactive placebo.The subject will orally consume the Vitamin D/placebo tablet 3 times a week for the 1st 8 weeks (while in hospital) and then once every other week for the last 8 weeks( during out-patient visits to the hospital).

The main study hypothesis is that Vitamin D supplementation helps patients with tuberculosis, who are on standard anti TB antibiotic therapy, get better faster.

DETAILED DESCRIPTION:
This is a double-blind, randomized, controlled clinical trial on the clinical efficacy and antimicrobial mechanisms of oral high dose vitamin D3 therapy three times weekly given for 8 weeks followed by the same vitamin D dose given every other week for a subsequent 8 weeks (n=129) versus placebo (n=129) in newly diagnosed Georgian patients with pulmonary TB.

The trial is also designed to obtain needed information on vitamin D status and general nutritional status in TB patients in Georgia, explore vitamin D regulation of the endogenous antimicrobial peptide cathelicidin/LL-37 in human tissues, and obtain hypothesis-generating data on the potential role of cathelicidin/LL-37 as a mechanism for the anti-mycobacterial effects of vitamin D in humans.

The potential study subjects will be identified and clinically monitored by clinical study coordinators after diagnosis by standard methods (compatible signs and symptoms, positive sputum AFB smear and culture, chest X-ray). Medical records of all patients with newly diagnosed tuberculosis registered for treatment at the NCTBLD in Tbilisi will be screened for eligibility for participation in the study. Written informed consent will be obtained from patients who met eligibility criteria and agreed to participate in the study prior to the subject undergoing any study-related procedure. Participation in study will involve a total of seven study visits (one baseline and six follow up visits.

TB patients will otherwise be conventionally treated with anti-TB drug regimens using the DOTS protocols: an initial 2 month in-hospital intensive phase with daily treatment with oral rifampicin, isoniazid, pyrazinamide and ethambutol, followed by an outpatient continuation phase for 4 months with rifampicin and isoniazid only, given 3 times per week. Given data that TB disease itself is associated with vitamin D depletion we will also recruit 80 otherwise healthy, adult family members of the pulmonary TB patients as a pilot substudy. Family members recruited will be those accompanying the TB patient to clinic.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is age > 18 years;
2. Patient has documented new case of smear-positive pulmonary TB;
3. Patient has received ≤ 1 week of anti-TB therapy;
4. The patient will receive anti-TB therapy in Tbilisi;
5. Patient has provided informed consent.

Exclusion Criteria:

1. Patient has had > 30 days of lifetime TB therapy;
2. Patient is currently pregnant or lactating;
3. Patient has a history of organ transplant;
4. Patient has a history of cancer in past 5 years (ineligibility criteria does not include non-melanoma skin cancer);
5. Patient has a history of seizures;
6. Patient has a history of hypercalcemia;
7. Patient has a history of hyperparathyroidism;
8. Patient has a history of sarcoidosis;
9. Patient has a history of nephrolithiasis (renal stones);
10. Patient has taken oral corticosteroids in the past 30 days;
11. Patient is currently using cytotoxic or immunosuppressive drugs;
12. Patient currently has significant renal dysfunction (defined as a serum creatinine of >250mmol/L);
13. Patient requires dialysis therapy;
14. Patient has a history of cirrhosis;
15. Patient is currently incarcerated;
16. Patient is not able to complete all study visits in at the NCTBLD in Tbilisi.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2009-07; Primary Completion 2012-09 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
The primary outcome for this intent-to-treat trial is the time to Mycobacterium tuberculosis sputum culture conversion to negative | Up to 16 weeks from therapy start date

SECONDARY OUTCOMES:
Sputum culture result (positive or negative) | 8 weeks after therapy start date

CONTACTS AND LOCATIONS:
Overall Officials: Thomas R Ziegler, MD, Principal Investigator — Emory University
Locations (1):
- National Center for tuberculosis and Lung diseases, Tbilisi, Georgia

REFERENCES:
- [Derived] Tukvadze N, Sanikidze E, Kipiani M, Hebbar G, Easley KA, Shenvi N, Kempker RR, Frediani JK, Mirtskhulava V, Alvarez JA, Lomtadze N, Vashakidze L, Hao L, Del Rio C, Tangpricha V, Blumberg HM, Ziegler TR. High-dose vitamin D3 in adults with pulmonary tuberculosis: a double-blind randomized controlled trial. Am J Clin Nutr. 2015 Nov;102(5):1059-69. doi: 10.3945/ajcn.115.113886. Epub 2015 Sep 23. PMID 26399865